CLINICAL TRIAL: NCT03850301
Title: An Experimental Medicine Study to Validate the 18 kiloDalton Translocator Protein (TSPO) as a Novel Neuroimmunodulatory Target in Multiple Sclerosis
Brief Title: Validation of the 18 kiloDalton Translocator Protein (TSPO) as a Novel Neuroimmunodulatory Target
Acronym: TSPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 17HH3814
Record Dates: First submitted 2019-02-12; First posted 2019-02-21 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — N-benzyl-N-ethyl-2-(7,8-dihydro-7-methyl-8-oxo-2-phenyl-9H-purin-9-yl)acetamide; etifoxine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The people who undertake the analysis of the blood test will be blind about whether the blood sample came from an MS patient or a healthy volunteer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etifoxine then XBD173 (Experimental)
  Interventions: Drug: XBD173; Drug: Etifoxine
- XBD173 then Etifoxine (Experimental)
  Interventions: Drug: XBD173; Drug: Etifoxine

INTERVENTIONS:
Drug: XBD173 — 7 days treatment
Drug: Etifoxine — 7 days treatment

SUMMARY:
In multiple sclerosis (MS) cells of the immune system attack the brain causing tissue damage. In secondary progressive MS (SPMS) these repeated immune attacks have stopped but despite this new damage continues to appear. TSPO is a protein found in the brain and cells of the immune system, whose levels increase during MS. The investigators would like to know whether drugs that bind TSPO could dampen the immune responses in patients with SPMS. The investigators will be testing two drugs that affect TSPO; etifoxine and XBD173. Subjects with SPMS will be recruited from neurology clinics at hospitals associated with Imperial College Healthcare NHS Trust. Healthy volunteers will also be recruited in order to provide a comparison to these patients. The volunteers recruited will be invited to the clinical research facility (CRF) at Hammersmith Hospital. The volunteers will take one of the two drugs every day for 7 days. The researchers will perform blood tests before the first dose and after the last dose to investigate the effects of the drugs, including the expression of genes and immune cell activity. This will allow the researchers to explore which of the two drugs produces the greatest changes in the amount of TSPO in the blood in MS patients relative to healthy controls.

DETAILED DESCRIPTION:
The 18 kiloDalton Translocator Protein (TSPO) is a mitochondrial protein highly expressed in myeloid cells. While the full range of its functions are unknown, preclinical and in vitro studies provide suggestive evidence that TSPO ligands alter TSPO protein function to bias monocytes/macrophages and microglia towards reparative phenotypes. XBD173 and etifoxine are two TSPO ligands and represent two distinct chemotypes. Etifoxine is a benzoxaine, licenced in France (although not the UK) for the treatment of anxiety. XBD173 (Emapunil) is a phenylpurine that has recently been investigated for the treatment of anxiety, but is not licensed.

The aim of this experimental medicine study is to test the hypothesis in humans that functional changes effected by TSPO can induce pro-inflammatory monocytes/macrophages and microglia to adopt a reparative phenotype. People with multiple sclerosis (MS) will be enrolled in this study because monocytes from MS patients have a chronic pro-inflammatory phenotype. Healthy volunteers (HVs) will also be enrolled to determine whether TSPO mediated effects are immune state dependant.

The primary objective of this study is to determine the effects of TSPO ligand binding on monocyte/macrophage phenotype in humans.

The secondary objectives are:

a To characterise immunological responses in blood plasma and in circulating immune cell subsets of healthy volunteers and people with SPMS after TSPO functional changes induced by challenge ligand binding.

b To explore the potential dependence of these pharmacodynamic responses on variation at rs6971 (a common polymorphism influencing ligand binding affinities in the TSPO protein) in the TSPO gene.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
2. Aged 35-65 years old
3. A female subject is eligible to participate if she is a) of non-childbearing potential, defined as pre-menopausal females with a documented tubal ligation or hysterectomy, or postmenopausal defined as 12 months of spontaneous amenorrhea or b) of childbearing potential but not pregnant (as determined by urinary pregnancy test on screening and on each study day) and willing to use one of the contraception methods listed below
4. Male subject must agree to use one of the contraception methods listed above.
5. Willing to abstain from alcohol for the duration of dosing.
6. Expanded Disability Status Scale (EDSS) >3.5 <6.5 (SPMS patients only)

Exclusion Criteria:

1. History of active neurological disease other than migraine or MS
2. Clinically meaningful abnormalities in routine bloods including:

   * eGFR < 60ml/min
   * Elevation of liver enzymes/bilirubin
   * Prolonged prothrombin time
   * Thrombocytopenia
3. Use of the following medications or therapies:

   * Immunosuppressive or immunomodulatory drugs within the last 6 months
   * Alemtuzumab or haematopeotic stem cell therapy
   * Central nervous system depressants (including opioid analgesics, barbiturates, sleeping pills, antihistamines, antipsychotics)
   * P450 CY3A4 inducers or inhibitors
   * oral contraceptives
   * oral anticoagulants or antiplatelet agents other than low dose aspirin
   * levothyroxine
4. Currently breastfeeding
5. Any clinical significant medical conditions that in the opinion of the investigator would compromise subjects' safety or compliance with study procedures.
6. History of any clinical condition which in the opinion of the principal investigator would compromise the scientific integrity of the study, such as some chronic systemic diseases affecting blood, liver or kidneys or endocrine system
7. Unwillingness or inability to follow the procedures outlined in the protocol
8. Subject is mentally or legally incapacitated
9. Contraindication to XBD173 use:

   • Hypersensitivity to the active substance or to any of the excipients
10. Contraindication to etifoxine use:

    * Myasthenia gravis
    * syndromes of glucose and galactose malabsorption or lactose deficiency

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Monocyte phenotye - Tissue necrosis factor-α | 7 days
  Plasma cytokine concentrations
Monocyte phenotye - Interferon-γ | 7 days
  Plasma cytokine concentrations
Monocyte phenotype - Interleukins- 1β | 7 days
  Plasma cytokine concentrations
Monocyte phenotype - Interleukins- 16 | 7 days
  Plasma cytokine concentrations
Monocyte phenotype - Interleukins- 17 | 7 days
  Plasma cytokine concentrations
Monocyte phenotype - Interleukins- 23 | 7 days
  Plasma cytokine concentrations
Immunomodulatory factor -Transforming growth factor-β | 7 days
  Transforming growth factor-β
Immunomodulatory factor - Interleukins -4 | 7 days
  Interleukins -4
Immunomodulatory factor - Interleukins - 10 | 7 days
  Interleukins - 10
Relative proportions of WBC subsets | 7 days
  Flow

SECONDARY OUTCOMES:
Monocyte phenotype - 'omic analyses | 7 days
  Genome, proteome, metabolome
Neurofilament | 7 days
  Plasma levels of neurofilament

CONTACTS AND LOCATIONS:
Overall Officials: Paul Matthews, PhD, Study Chair — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided